CLINICAL TRIAL: NCT04805840
Title: Comparison of Screening for SARS-CoV-2 (COVID-19) in a Low Prevalence Setting Using Serial Antigen Testing Versus Serial Molecular (PCR) Testing
Brief Title: Sensitivity of Frequent SARS-CoV-2 (COVID-19) Rapid Antigen Testing Regimen
Status: Terminated | Type: Observational
Why Stopped: Difficulty with recruitment.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAT5233
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: COVID-19; COVID; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: CoV-SCAN rapid COVID-19 antigen test — SARS-CoV-2 rapid antigen screening test

SUMMARY:
This study aims to assess how an at-home COVID-19 frequent testing regimen using the CoV-SCAN test kit and a paired phone application to help interpret the test result compares to once-a-week or three-times-a-week polymerase chain reaction (PCR) (molecular) testing to identify a SARS-CoV-2 infection.

Employees and cast members at Media and Entertainment Company and its affiliates will be recruited to test whether frequent use of CoV-SCAN will perform as well or better than weekly molecular testing and at least as well as three-times-a-week molecular testing.

DETAILED DESCRIPTION:
Antigen tests are simple to perform, have a rapid turn-around time of 15-30 minutes, and a lower cost than molecular tests. Because antigen tests do not incorporate an amplification step, they are intrinsically less sensitive than PCR molecular tests. Nevertheless, several investigators have examined the feasibility of screening populations of individuals in a low SARS-CoV-2 infection prevalence situation, such as the workplace or schools, with rapid antigen tests in place of the molecular tests. Using viral kinetics, knowledge of what level of viral load is required for transmission of culture-competent virus, test sensitivity and modeling, they have come to the conclusion that more frequent testing with a test with lower sensitivity that has a quick turn-around time is better than a test with high sensitivity with a longer turn-around time. Therefore, the goal of this study is to test the hypothesis that frequent testing with a relatively sensitive lateral flow antigen test performed at home using self-collected anterior nasal swabs will be superior to once a week or less PCR testing and non-inferior to three times a week PCR testing in an employment screening setting with a relatively low incidence of new SARS-CoV-2 infections. This study aims to assess how an at-home COVID-19 frequent testing regimen using a Rapid Antigen Screening Test (RAST) and a phone application to help interpret the test result compares to once-a-week or three-times-a-week PCR (molecular) testing to identify a SARS-CoV-2 infection. We expect to recruit up to 4,400 employees and cast members of Media and Entertainment Company and its affiliates to test whether frequent use of the RAST will perform as well or better than weekly molecular testing and at least as well as three-times-a-week molecular testing. Recruitment and the study will continue until at least 31 or at most 148 true positive SARS-CoV-2 molecular results are reached.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Have a smartphone;
* Understand and read English;
* Will be on one production location for at least three weeks following enrollment to the study;
* Will be willing to be contacted by the Study Coordinator after leaving one production location to facilitate continued access to weekly molecular testing;

Exclusion Criteria:

* Have received any dose of COVID-19 vaccination;
* Have been diagnosed with COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees and cast members of a Media and Entertainment Company
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Sensitivity of CoV-SCAN daily testing regimen | Baseline to 21 days
  To compare the sensitivity (the percentage of people with the disease who test positive) of the rapid antigen testing regimen to the gold standard PCR testing regimen
Specificity of CoV-SCAN daily testing regimen | Baseline to 21 days
  To compare the specificity (the ability of the test to correctly identify those without the disease) of the rapid antigen testing regimen to the gold standard PCR testing regimen

SECONDARY OUTCOMES:
Time from CoV-SCAN positive to PCR positive result | Baseline to 21 days
  To compare time to diagnosis with the rapid antigen testing regimen to the gold standard PCR testing regimen

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine Meyers, DrPH, MS, MPP, Principal Investigator — Assistant Professor
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States